CLINICAL TRIAL: NCT02975128
Title: Minimal Invasive Breast Cancer Excision Using the Breast Lesion Excision System Under Ultrasound Guidance
Acronym: BLES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Needle production stopped
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL58040.091.16
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breastcancer
Keywords: Minimal invasive; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: BLES system and conventional lumpectomy

INTERVENTIONS:
Device: BLES system and conventional lumpectomy — Each patient undergoes the same procedure. Under general anaesthesia for the normal surgical procedure, the tumor is first removed using the BLES system under US guidance. Next, the normal surgical procedure is performed, excising the BLES excision cavity and a ≥ 1cm margin of surrounding tissue, also guided by the US appearance after the BLES procedure.

SUMMARY:
This study will assess whether it is feasible to remove small breast cancers completely using the Breast Lesion Excision System under Ultrasound guidance.

DETAILED DESCRIPTION:
Rationale: In the Netherlands, ≥7000 women are operated for small breast cancers yearly. In this study, we will evaluate under which conditions it is possible to excise small breast cancers using the Breast Lesion Excision System (BLES) under ultrasound (US) guidance. When successful, this will allow ambulatory treatment of women with small breast cancers, improving the cosmetic outcome and quality of life.

Objective: Our study aim is to assess whether it is feasible to remove small breast cancers completely using the BLES system under US guidance.

Study design: This is a multi-centre, translational clinical phase II study in 125 women with cancers ≤1.5 cm based upon US measurements, and without mammographic evidence of more extensive disease (e.g. microcalcifications).

Study population: Women with cancers ≤1.5 cm based upon US measurements, if there is no mammographic evidence of more extensive disease (e.g. microcalcifications or extensive architectural distortion), and the tumor lies ≥6 mm away from the dermis, nipple or pectoral muscle, are eligible for this study.

Intervention: In 125 women with cancers ≤1.5 cm based upon US measurements, and without mammographic evidence of more extensive disease (e.g. microcalcifications), we will conduct additional preoperative breast MRI to ascertain lesion size, after informed consent has been obtained. If the lesion is confirmed ≤1.5 cm on MRI and lying ≥6 mm away from the dermis, nipple and pectoral muscle, the patient is eligible. Moreover, patients will be asked to fill out the questionnaire, detailing their risk profile and comorbidity index.

Under general anaesthesia for the normal surgical procedure, the tumor is first removed using the BLES system under US guidance, through a small skin incision (<1 cm). Next, the normal surgical procedure is performed, excising the BLES excision cavity and a ≥ 1cm margin of surrounding tissue, also guided by the US appearance after the BLES procedure. Margin assessment will be performed separately for the BLES excision and the surgical specimen of the surrounding tissue.

Main study parameters/endpoints: Main endpoint of the study is the frequency of successful complete tumor excision by the BLES system, where successful is defined as 'having tumor free margins, and no residual (in situ) cancer in the surgical specimen'.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Our approach allows to test the feasibility of this highly innovating approach to remove breast cancer, with minimal negative effects or possible complications.

While there is no direct benefit nor detrimental effect from this study to the patients participating, the study has large implications for many women, as breast cancer remains the most common cancer in women, and due to screening, most cancers are small. Further reduction of the impact of local treatment is still desired as the psychosocial and somatic effects of breast deformation can be substantial.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 19 years or older
* US visible breast cancer with maximum diameter of 15 mm on US
* Histologically proven invasive breast cancer
* Willing and able to undergo preoperative breast MRI
* Able to provide informed consent

Exclusion Criteria:

* Poor US visibility of the breast cancer
* Breast cancer closer than 6 mm to the dermis, nipple or pectoral muscle.
* Contra-indications to breast MRI or intravenous contrast administration
* Contra-indications for the use of diathermia
* Unable to provide informed consent
* Patients with breast implants
* Patients with implanted electronics
* Pregnancy
* Neoadjuvant chemotherapy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of successful complete tumor excision by the BLES system. | Through study completion, an average of two months
  Successful is defined as 'having tumor free margins, and no residual (in situ) cancer in the surgical specimen'.

SECONDARY OUTCOMES:
Quality of the margin evaluation of the biopsy specimen and the eventual surgical specimen. | Through study completion, an average of two months
In biopsy specimen in which the margin is not completely tumor free, but the Dutch criterion for successful surgery is met (no more than focal (4 mm) margin involvement), we will specifically analyse the residual tumor burden in the surgical excision. | Through study completion, an average of two months
Assess in retrospect whether we can predict successful tumor extraction based upon other factors than tumor size alone. | 2 years
  Parameters categorized in:
  * Patient related variables obtained from a questionnaire
  * Lesion related variables
  * Imaging features
  * Surgical features
  * Histopathological and molecular features from the core biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ritse Mann, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland

REFERENCES:
- [Background] Allen SD, Nerurkar A, Della Rovere GU. The breast lesion excision system (BLES): a novel technique in the diagnostic and therapeutic management of small indeterminate breast lesions? Eur Radiol. 2011 May;21(5):919-24. doi: 10.1007/s00330-010-2000-7. Epub 2011 Jan 15. PMID 21240608
- [Background] Sie A, Bryan DC, Gaines V, Killebrew LK, Kim CH, Morrison CC, Poller WR, Romilly AP, Schilling K, Sung JH. Multicenter evaluation of the breast lesion excision system, a percutaneous, vacuum-assisted, intact-specimen breast biopsy device. Cancer. 2006 Sep 1;107(5):945-9. doi: 10.1002/cncr.22090. PMID 16874817
- [Background] Medjhoul A, Canale S, Mathieu MC, Uzan C, Garbay JR, Dromain C, Balleyguier C. Breast lesion excision sample (BLES biopsy) combining stereotactic biopsy and radiofrequency: is it a safe and accurate procedure in case of BIRADS 4 and 5 breast lesions? Breast J. 2013 Nov-Dec;19(6):590-4. doi: 10.1111/tbj.12184. Epub 2013 Sep 19. PMID 24102869
- [Background] Allen SD, Osin P, Nerurkar A. The radiological excision of high risk and malignant lesions using the INTACT breast lesion excision system. A case series with an imaging follow up of at least 5 years. Eur J Surg Oncol. 2014 Jul;40(7):824-9. doi: 10.1016/j.ejso.2014.03.022. Epub 2014 Apr 2. PMID 24742589